CLINICAL TRIAL: NCT02772679
Title: A Phase 1 Trial of CD4+CD127lo/-CD25+ Polyclonal Treg Adoptive Immunotherapy With Interleukin-2 for the Treatment of Type 1 Diabetes
Brief Title: T1DM Immunotherapy Using Polyclonal Tregs + IL-2
Acronym: TILT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey Bluestone (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Bluestone, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-19632
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes; Treg; Proluekin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- PolyTregs+IL-2 (Experimental): Patients with type 1 diabetes mellitus will receive ex vivo expanded human autologous polyclonal regulatory T cells plus IL-2
  Interventions: Biological: PolyTregs+IL-2

INTERVENTIONS:
Biological: PolyTregs+IL-2 — PolyTregs will be infused into the patient in a single infusion. The first cohort will receive 3 x10^6 cells. The second cohort will receive 20x10^6 cells. Following the day 0 infusion of polyclonal Tregs, subjects will receive two 5-day courses of IL-2 (1 x 106 IU daily), the first on days 3-7 and the second on days 38-42. Administration of the second course of IL-2 may be delayed or withheld depending on threshold criteria for peripheral blood Treg frequencies and MMTT-stimulated C-peptide levels determined on day 28.

SUMMARY:
The purpose of this study is to assess the safety of Tregs + IL-2 and survival of Tregs in patients with recent onset T1DM who receive infusions of autologous Tregs + IL-2.

DETAILED DESCRIPTION:
The investigators hypothesize that ex vivo expanded human autologous CD4+CD127lo/-CD25+ polyclonal regulatory T cells (Polyclonal Tregs) plus Interleukin-2 (IL-2) administered to patients with Type 1 Diabetes Mellitus (T1DM) will be safe and biologically active. A Phase I trial with this cellular therapy plus IL-2 will lead the way for Phase II trials that test for efficacy based on preservation of C-peptide, reduced exogenous insulin requirements and improved glycemic control.

This is a Phase I safety/dosing study of Polyclonal Tregs + IL-2 in patients with T1DM.

The Tregs will be expanded using an established protocol utilizing anti-CD3/anti-CD28 beads plus IL-2. The study will involve 2 dosing cohorts of 6-8 T1DM patients each. The primary objective of this study is to assess the safety of Tregs + IL-2 and survival of Tregs in patients with recent onset T1DM who receive infusions of autologous Tregs + IL-2. The study will also assess potential effects of Tregs on beta cell function and the autoimmune response.

Subjects will receive Polyclonal Tregs at doses of 3 or 20x10^6 cells/kg. The dose of Tregs is selected based on a combination of considerations of manufacturing capacity, a predicted efficacious dose, and the available safety data of the Treg product currently in clinical trials. The IL-2 dose will be 1 x10^6 IU subcutaneously, given daily for 5 consecutive days at the completion of the cell infusion and again after 1 month. This dose is based on recent studies from Klatzmann et al. in T1DM, where the dose was found to be effective in a selective Treg expansion, well tolerated, and without an acute decline in beta cell function (Rosenzwajg et al., 2015).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of T1DM within >3 and <24 months of day 0 according to the American Diabetes Association standard criteria.
2. 18 to 45 years of age on day of screening visit.
3. Positive for at least one islet cell autoantibody (glutamate decarboxylase; insulin, if obtained within 10 days of the onset of insulin therapy; ICA 512-antibody; and/or ZnT8).
4. Peak stimulated C-peptide level >0.2 pmol/mL (0.6 ng/ml) following an MMTT.
5. Weight of >= 40 kg and <=90.7kg
6. Adequate venous access to support a blood draw of 5 mls/kg up to maximum of 400 ml whole blood and later infusion of investigational therapy

Exclusion Criteria:

1. Hemoglobin <10.0 g/dL; leukocytes <3,000/μL; neutrophils <1,500/μL; lymphocytes <800μL; platelets <100,000/μL
2. Any sign of significant chronic active infection (e.g., hepatitis, tuberculosis, EBV, or CMV), or screening laboratory evidence consistent with a significant chronic active infection (such as positive for HIV, PPD, or HBsAg).
3. Anticipated ongoing use of diabetes medications other than insulin that affect glucose homeostasis, such as metformin, sulfonylureas, thiazolidinediones, glucagon-like peptide 1 (GLP-1) mimetics, dipeptidyl peptidase IV (DPP-IV) inhibitors, SGLT2 inhibitors, or amylin.
4. Chronic use of systemic glucocorticoids or other immunosuppressive agents, or biologic immunomodulators within 6 months prior to study entry. Specifically, subjects who have received over 7 days of treatment with 7.5 mg of prednisone (or the equivalent) within 6 months prior to study entry will be excluded.
5. History of malignancy (including squamous cell carcinoma of the skin or cervix) except adequately treated basal cell carcinoma
6. Pregnant or breastfeeding women, or any female who is unwilling to use a reliable and effective form of contraception for 1 year after Treg +/- IL-2 dosing, and any male who is unwilling to use a reliable and effective form of contraception for 3 months after Treg +/- IL-2 dosing
7. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results.
8. Patients who are unwilling to agree to not participate in another clinical trial, which in the opinion of the investigator may confound the results of this study, for at least 1 year following Treg infusion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08; Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Adverse events | up to 3 years
  Adverse events of special interest: including infections, malignancies, safety of Treg infusions, and local and systemic reactions to IL-2.
Survival of Tregs | up to 3 years
  Comparison of the survival of graded doses of Tregs and IL-2. Calculating the half-life of infused deuterium-labeled Tregs in peripheral circulation will be used to assess the survival of Tregs.

SECONDARY OUTCOMES:
C-peptide response | up to 3 years
  Change in beta cell function over time, as assessed by change in C-peptide area under curve in response to serial mixed meal tolerance tests. Analysis will include a comparison to recent data available from TrialNet placebo treated subjects.
Insulin use | up to 3 years
  Insulin use in units per kilogram body weight per day
HbA1c levels | up to 3 years
Severe hypoglycemic events | up to 3 years
  Severe hypoglycemic events as defined by the inability to selftreat and/or the requirement for glucagon injection
Proportion of subjects who achieve at least a 13-week reduction in insulin dose to < 0.5 units/kg in each treatment arm | up to 3 years
Analysis of the effects of IL-2 on Treg kinetics and phenotype | up to 3 years
Levels of unmethylated insulin DNA (assay of beta cell death) | up to 3 years
Analysis of autoantibodies, enumeration and phenotypes islet antigen tetramer+ CD8, intracellular cytokine staining of T cells, serum proteomics, cytokines, and Treg phenotyping and functional assays | up to 3 years
Analysis of general immune response as assessed by, for example, viral tetramer+ CD8 cells and effects of Treg infusions on peripheral blood cells measured by flow cytometry including T cell subsets, B cells and other innate cell subsets | up to 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Francisco Medical Center, San Francisco, California
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chatenoud L, Bluestone JA. CD3-specific antibodies: a portal to the treatment of autoimmunity. Nat Rev Immunol. 2007 Aug;7(8):622-32. doi: 10.1038/nri2134. Epub 2007 Jul 20. PMID 17641665
- [Background] Ahmadzadeh M, Rosenberg SA. IL-2 administration increases CD4+ CD25(hi) Foxp3+ regulatory T cells in cancer patients. Blood. 2006 Mar 15;107(6):2409-14. doi: 10.1182/blood-2005-06-2399. Epub 2005 Nov 22. PMID 16304057
- [Background] Ash S, Yarkoni S, Askenasy N. Lymphopenia is detrimental to therapeutic approaches to type 1 diabetes using regulatory T cells. Immunol Res. 2014 Jan;58(1):101-5. doi: 10.1007/s12026-013-8476-x. PMID 24371009
- [Background] Atkins MB. Interleukin-2: clinical applications. Semin Oncol. 2002 Jun;29(3 Suppl 7):12-7. doi: 10.1053/sonc.2002.33077. PMID 12068383
- [Background] Bailey-Bucktrout SL, Martinez-Llordella M, Zhou X, Anthony B, Rosenthal W, Luche H, Fehling HJ, Bluestone JA. Self-antigen-driven activation induces instability of regulatory T cells during an inflammatory autoimmune response. Immunity. 2013 Nov 14;39(5):949-62. doi: 10.1016/j.immuni.2013.10.016. PMID 24238343
- [Background] Bayer AL, Pugliese A, Malek TR. The IL-2/IL-2R system: from basic science to therapeutic applications to enhance immune regulation. Immunol Res. 2013 Dec;57(1-3):197-209. doi: 10.1007/s12026-013-8452-5. PMID 24214027
- [Background] Bluestone JA. Regulatory T-cell therapy: is it ready for the clinic? Nat Rev Immunol. 2005 Apr;5(4):343-9. doi: 10.1038/nri1574. PMID 15775994
- [Background] Buckner JH. Mechanisms of impaired regulation by CD4(+)CD25(+)FOXP3(+) regulatory T cells in human autoimmune diseases. Nat Rev Immunol. 2010 Dec;10(12):849-59. doi: 10.1038/nri2889. PMID 21107346
- [Background] Castela E, Le Duff F, Butori C, Ticchioni M, Hofman P, Bahadoran P, Lacour JP, Passeron T. Effects of low-dose recombinant interleukin 2 to promote T-regulatory cells in alopecia areata. JAMA Dermatol. 2014 Jul;150(7):748-51. doi: 10.1001/jamadermatol.2014.504. PMID 24872229
- [Background] Churlaud G, Jimenez V, Ruberte J, Amadoudji Zin M, Fourcade G, Gottrand G, Casana E, Lambrecht B, Bellier B, Piaggio E, Bosch F, Klatzmann D. Sustained stimulation and expansion of Tregs by IL2 control autoimmunity without impairing immune responses to infection, vaccination and cancer. Clin Immunol. 2014 Apr;151(2):114-26. doi: 10.1016/j.clim.2014.02.003. Epub 2014 Feb 19. PMID 24576619
- [Background] Couri CE, Oliveira MC, Stracieri AB, Moraes DA, Pieroni F, Barros GM, Madeira MI, Malmegrim KC, Foss-Freitas MC, Simoes BP, Martinez EZ, Foss MC, Burt RK, Voltarelli JC. C-peptide levels and insulin independence following autologous nonmyeloablative hematopoietic stem cell transplantation in newly diagnosed type 1 diabetes mellitus. JAMA. 2009 Apr 15;301(15):1573-9. doi: 10.1001/jama.2009.470. PMID 19366777
- [Background] Diaz-de-Durana Y, Lau J, Knee D, Filippi C, Londei M, McNamara P, Nasoff M, DiDonato M, Glynne R, Herman AE. IL-2 immunotherapy reveals potential for innate beta cell regeneration in the non-obese diabetic mouse model of autoimmune diabetes. PLoS One. 2013 Oct 24;8(10):e78483. doi: 10.1371/journal.pone.0078483. eCollection 2013. PMID 24205242
- [Background] Dirice E, Kahraman S, Jiang W, El Ouaamari A, De Jesus DF, Teo AK, Hu J, Kawamori D, Gaglia JL, Mathis D, Kulkarni RN. Soluble factors secreted by T cells promote beta-cell proliferation. Diabetes. 2014 Jan;63(1):188-202. doi: 10.2337/db13-0204. Epub 2013 Oct 2. PMID 24089508
- [Background] Garg G, Tyler JR, Yang JH, Cutler AJ, Downes K, Pekalski M, Bell GL, Nutland S, Peakman M, Todd JA, Wicker LS, Tree TI. Type 1 diabetes-associated IL2RA variation lowers IL-2 signaling and contributes to diminished CD4+CD25+ regulatory T cell function. J Immunol. 2012 May 1;188(9):4644-53. doi: 10.4049/jimmunol.1100272. Epub 2012 Mar 28. PMID 22461703
- [Background] Grinberg-Bleyer Y, Baeyens A, You S, Elhage R, Fourcade G, Gregoire S, Cagnard N, Carpentier W, Tang Q, Bluestone J, Chatenoud L, Klatzmann D, Salomon BL, Piaggio E. IL-2 reverses established type 1 diabetes in NOD mice by a local effect on pancreatic regulatory T cells. J Exp Med. 2010 Aug 30;207(9):1871-8. doi: 10.1084/jem.20100209. Epub 2010 Aug 2. PMID 20679400
- [Background] Hartemann A, Bensimon G, Payan CA, Jacqueminet S, Bourron O, Nicolas N, Fonfrede M, Rosenzwajg M, Bernard C, Klatzmann D. Low-dose interleukin 2 in patients with type 1 diabetes: a phase 1/2 randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2013 Dec;1(4):295-305. doi: 10.1016/S2213-8587(13)70113-X. Epub 2013 Oct 8. PMID 24622415
- [Background] Johnson MC, Garland AL, Nicolson SC, Li C, Samulski RJ, Wang B, Tisch R. beta-cell-specific IL-2 therapy increases islet Foxp3+Treg and suppresses type 1 diabetes in NOD mice. Diabetes. 2013 Nov;62(11):3775-84. doi: 10.2337/db13-0669. Epub 2013 Jul 24. PMID 23884888
- [Background] Liu R, Zhou Q, La Cava A, Campagnolo DI, Van Kaer L, Shi FD. Expansion of regulatory T cells via IL-2/anti-IL-2 mAb complexes suppresses experimental myasthenia. Eur J Immunol. 2010 Jun;40(6):1577-89. doi: 10.1002/eji.200939792. PMID 20352624
- [Background] Macallan DC, Asquith B, Zhang Y, de Lara C, Ghattas H, Defoiche J, Beverley PC. Measurement of proliferation and disappearance of rapid turnover cell populations in human studies using deuterium-labeled glucose. Nat Protoc. 2009;4(9):1313-27. doi: 10.1038/nprot.2009.117. Epub 2009 Aug 20. PMID 19696750
- [Background] Malek TR, Pugliese A. Low-dose IL-2 as a therapeutic agent for tolerance induction. Immunotherapy. 2011 Nov;3(11):1281-4. doi: 10.2217/imt.11.120. No abstract available. PMID 22053878
- [Background] Marek-Trzonkowska N, Mysliwiec M, Dobyszuk A, Grabowska M, Derkowska I, Juscinska J, Owczuk R, Szadkowska A, Witkowski P, Mlynarski W, Jarosz-Chobot P, Bossowski A, Siebert J, Trzonkowski P. Therapy of type 1 diabetes with CD4(+)CD25(high)CD127-regulatory T cells prolongs survival of pancreatic islets - results of one year follow-up. Clin Immunol. 2014 Jul;153(1):23-30. doi: 10.1016/j.clim.2014.03.016. Epub 2014 Apr 1. PMID 24704576
- [Background] Marek-Trzonkowska N, Mysliwiec M, Dobyszuk A, Grabowska M, Techmanska I, Juscinska J, Wujtewicz MA, Witkowski P, Mlynarski W, Balcerska A, Mysliwska J, Trzonkowski P. Administration of CD4+CD25highCD127- regulatory T cells preserves beta-cell function in type 1 diabetes in children. Diabetes Care. 2012 Sep;35(9):1817-20. doi: 10.2337/dc12-0038. Epub 2012 Jun 20. PMID 22723342
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Monti P, Heninger AK, Bonifacio E. Differentiation, expansion, and homeostasis of autoreactive T cells in type 1 diabetes mellitus. Curr Diab Rep. 2009 Apr;9(2):113-8. doi: 10.1007/s11892-009-0020-y. PMID 19323955
- [Background] Putnam AL, Brusko TM, Lee MR, Liu W, Szot GL, Ghosh T, Atkinson MA, Bluestone JA. Expansion of human regulatory T-cells from patients with type 1 diabetes. Diabetes. 2009 Mar;58(3):652-62. doi: 10.2337/db08-1168. Epub 2008 Dec 15. PMID 19074986
- [Background] Salomon B, Bluestone JA. Complexities of CD28/B7: CTLA-4 costimulatory pathways in autoimmunity and transplantation. Annu Rev Immunol. 2001;19:225-52. doi: 10.1146/annurev.immunol.19.1.225. PMID 11244036
- [Background] Sitrin J, Ring A, Garcia KC, Benoist C, Mathis D. Regulatory T cells control NK cells in an insulitic lesion by depriving them of IL-2. J Exp Med. 2013 Jun 3;210(6):1153-65. doi: 10.1084/jem.20122248. Epub 2013 May 6. PMID 23650440
- [Background] Tang Q, Adams JY, Penaranda C, Melli K, Piaggio E, Sgouroudis E, Piccirillo CA, Salomon BL, Bluestone JA. Central role of defective interleukin-2 production in the triggering of islet autoimmune destruction. Immunity. 2008 May;28(5):687-97. doi: 10.1016/j.immuni.2008.03.016. Epub 2008 May 8. PMID 18468463
- [Background] Tang Q, Bluestone JA. Regulatory T-cell physiology and application to treat autoimmunity. Immunol Rev. 2006 Aug;212:217-37. doi: 10.1111/j.0105-2896.2006.00421.x. PMID 16903917
- [Background] Tang Q, Bluestone JA. The Foxp3+ regulatory T cell: a jack of all trades, master of regulation. Nat Immunol. 2008 Mar;9(3):239-44. doi: 10.1038/ni1572. PMID 18285775
- [Background] Tang Q, Boden EK, Henriksen KJ, Bour-Jordan H, Bi M, Bluestone JA. Distinct roles of CTLA-4 and TGF-beta in CD4+CD25+ regulatory T cell function. Eur J Immunol. 2004 Nov;34(11):2996-3005. doi: 10.1002/eji.200425143. PMID 15468055
- [Background] Tang Q, Henriksen KJ, Bi M, Finger EB, Szot G, Ye J, Masteller EL, McDevitt H, Bonyhadi M, Bluestone JA. In vitro-expanded antigen-specific regulatory T cells suppress autoimmune diabetes. J Exp Med. 2004 Jun 7;199(11):1455-65. doi: 10.1084/jem.20040139. PMID 15184499
- [Background] Waldron-Lynch F, Kareclas P, Irons K, Walker NM, Mander A, Wicker LS, Todd JA, Bond S. Rationale and study design of the Adaptive study of IL-2 dose on regulatory T cells in type 1 diabetes (DILT1D): a non-randomised, open label, adaptive dose finding trial. BMJ Open. 2014 Jun 4;4(6):e005559. doi: 10.1136/bmjopen-2014-005559. PMID 24898091
- [Background] Bluestone JA, Buckner JH, Fitch M, Gitelman SE, Gupta S, Hellerstein MK, Herold KC, Lares A, Lee MR, Li K, Liu W, Long SA, Masiello LM, Nguyen V, Putnam AL, Rieck M, Sayre PH, Tang Q. Type 1 diabetes immunotherapy using polyclonal regulatory T cells. Sci Transl Med. 2015 Nov 25;7(315):315ra189. doi: 10.1126/scitranslmed.aad4134. PMID 26606968
- [Derived] Dong S, Hiam-Galvez KJ, Mowery CT, Herold KC, Gitelman SE, Esensten JH, Liu W, Lares AP, Leinbach AS, Lee M, Nguyen V, Tamaki SJ, Tamaki W, Tamaki CM, Mehdizadeh M, Putnam AL, Spitzer MH, Ye CJ, Tang Q, Bluestone JA. The effect of low-dose IL-2 and Treg adoptive cell therapy in patients with type 1 diabetes. JCI Insight. 2021 Sep 22;6(18):e147474. doi: 10.1172/jci.insight.147474. PMID 34324441